CLINICAL TRIAL: NCT01896193
Title: A Phase 3b, Multicenter, Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of Sofosbuvir Plus Ribavirin in Treatment-Naïve Adults With Genotype 1 and 3 Chronic HCV Infection.
Brief Title: Safety and Efficacy Study of Sofosbuvir Plus Ribavirin in Treatment-Naive Adults With Genotype 1 and 3 Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0119
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOF+RBV 16 Weeks (Experimental): SOF+RBV for 16 weeks
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (Experimental): SOF+RBV for 24 weeks
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; PSI-7977; GS-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose using weight-based dosing (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir plus ribavirin administered for 16 weeks and 24 weeks in participants with chronic genotype 1 (GT1) or genotype 3 (GT3) hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed chronic genotype 1 or 3 HCV infection
* HCV treatment-naive
* Individuals will have cirrhosis status assessment; liver biopsy may be required.
* Screening laboratory values within predefined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Contraindication to ribavirin therapy
* Excessive alcohol ingestion as defined by protocol
* History of solid organ transplantation
* Current or prior history of clinical hepatic decompensation
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment, or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kersey, MSc, Study Director — Gilead Sciences
Locations (16):
- Russia (16):
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Central Scientific and Research Institute of Epidemiology of Rospotrebnadzor, Moscow
  - Central Scientific Research Institution of Gastroenterology of Moscow Healthcare Department, Moscow
  - City Clinical Hospital 24, Moscow
  - Clinical Diagnostics and Research Center of Federal Bedgetary Institution, Moscow
  - Infectious Clinical Hospital No. 1, Moscow
  - Institute of Nutrition of Academy of Sciences, Moscow
  - Institution of Healthcare of Sverdlovsk Region, Moscow
  - Institution of High Professional Education First Moscow State Medical University, Moscow
  - Institution of Tumen Region, Moscow
  - Krasnoyarsk Regional Center for Prevention and Control of AIDS and Infectious Diseases, Moscow
  - Scientific Research Institution of Emergency Care n.a. N.V. Sclifosovskiy of Moscow, Moscow
  - Stavropol State Medical University of Ministry of Healthcare, Moscow
  - Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Saint-Petersburg Center for Prevention and Control of AIDS and Infectious Diseases, Saint Petersburg
  - Medical Company Hepatolog, Samara

REFERENCES:
- [Derived] Isakov V, Zhdanov K, Kersey K, Svarovskaia E, Massetto B, Zhu Y, Knox SJ, Bakulin I, Chulanov V. Efficacy of sofosbuvir plus ribavirin in treatment-naive patients with genotype-1 and -3 HCV infection: results from a Russian Phase IIIb study. Antivir Ther. 2016;21(8):671-678. doi: 10.3851/IMP3065. Epub 2016 Jul 4. PMID 27376706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 16 study sites in Russia. The first participant was screened on 06 June 2013. The last study visit occurred on 27 July 2014.
Pre-assignment Details: 139 participants were screened.
Groups:
- SOF+RBV 16 Weeks: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 16 weeks
- SOF+RBV 24 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Started | 62 | 65
Completed | 41 | 53
Not Completed | 21 | 12
Not completed — Lack of Efficacy | 20 | 11
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- SOF+RBV 16 Weeks, GT1: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 16 weeks (genotype 1)
- SOF+RBV 24 Weeks, GT1: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (genotype 1)
- SOF+RBV 16 Weeks, GT3: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 16 weeks (genotype 3)
- SOF+RBV 24 Weeks, GT3: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (genotype 3)
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3 | Total
Number analyzed (Participants) | 32 | 34 | 30 | 31 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.8) | 42 (9.8) | 38 (8.2) | 40 (9.6) | 40 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 11 | 12 | 60
  Male | 13 | 16 | 19 | 19 | 67
Race/Ethnicity, Customized [Number; unit: participants]
  White | 32 | 34 | 30 | 31 | 127
Cirrhosis Status [Number; unit: participants]
  No | 28 | 28 | 23 | 26 | 105
  Yes | 4 | 6 | 6 | 5 | 21
  Missing | 0 | 0 | 1 | 0 | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 10 | 6 | 12 | 15 | 43
    CT | 19 | 23 | 16 | 15 | 73
    TT | 3 | 5 | 2 | 1 | 11
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.60) | 6.1 (0.60) | 6.2 (0.81) | 6.2 (0.77) | 6.2 (0.69)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 12 | 11 | 10 | 10 | 43
  ≥ 800,000 IU/mL | 20 | 23 | 20 | 21 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 1 or 3 HCV infection who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3
Number analyzed (Participants) | 32 | 34 | 30 | 31
percentage of participants | 50.0 | 76.5 | 86.7 | 90.3

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants permanently discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3
Number analyzed (Participants) | 32 | 34 | 30 | 31
percentage of participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3
Number analyzed (Participants) | 32 | 34 | 30 | 31
percentage of participants
  SVR4 | 53.1 | 76.5 | 90.0 | 90.3
  SVR24 | 46.9 | 76.5 | 86.7 | 90.3

4. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3
Number analyzed (Participants) | 32 | 34 | 30 | 31
percentage of participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Virologic Relapse
Description: Virologic relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 16 Weeks, GT1 | SOF+RBV 24 Weeks, GT1 | SOF+RBV 16 Weeks, GT3 | SOF+RBV 24 Weeks, GT3
Number analyzed (Participants) | 32 | 34 | 30 | 31
percentage of participants | 50.0 | 23.5 | 13.3 | 9.7

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- SOF+RBV 16 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 16 weeks
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 1/62 | 1/65
Other Adverse Events (participants affected / at risk) | 16/62 | 21/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 16 Weeks (N=62) | SOF+RBV 24 Weeks (N=65)
Pneumonia (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 16 Weeks (N=62) | SOF+RBV 24 Weeks (N=65)
Asthenia (General disorders) | 7 | 4
Fatigue (General disorders) | 2 | 4
Respiratory tract infection viral (Infections and infestations) | 3 | 5
Headache (Nervous system disorders) | 5 | 10
Insomnia (Psychiatric disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years